CLINICAL TRIAL: NCT03561662
Title: The Effect of Soya Foods on Cognitive Function and Menopausal Symptoms in Postmenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Alpro Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UREC/15/0025
Record Dates: First submitted 2018-05-02; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Menopause
Keywords: soya; menopause; cognitive function; isoflavones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low isoflavone (Active Comparator): Alpro soya drinks containing 10 mg isoflavones per day
  Interventions: Dietary Supplement: Alpro soya drinks
- Medium isoflavone (Active Comparator): Alpro soya drinks containing 35 mg isoflavones per day
  Interventions: Dietary Supplement: Alpro soya drinks
- High isoflavone (Active Comparator): Alpro soya drinks containing 60 mg isoflavones per day
  Interventions: Dietary Supplement: Alpro soya drinks

INTERVENTIONS:
Dietary Supplement: Alpro soya drinks — 12 weeks

SUMMARY:
Participants will be randomly assigned to one of three treatment groups to receive soyafoods (Alpro drinks) providing a low (<10 mg), medium (35mg) or high-dose (60 mg) of isoflavones daily for a period of 12 weeks. The group receiving <10mg isoflavones daily will serve as a low-dose control group. Women will be asked to avoid consuming any additional soya foods during the study.

Dietary intake will be assessed at baseline using the validated food frequency questionnaire a 4 day food diary will be completed at baseline and post-intervention. Weight and height will be measured and a general health & lifestyle questionnaire will also be completed by participants at baseline. Cognitive function will be assessed at baseline and post-intervention using the well validated and widely used computerised test battery system. Menopausal symptoms, quality of life, mood, stress and coping will also be assessed.

Plasma concentrations of the soya isoflavones genistein and daidzein will be measured to assess compliance. Circulating concentrations of equol (a daidzein metabolite), will also be measured to investigate associations between equol and cognition and menopausal symptoms as a potential mechanism for the efficacy of soya.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy
* within 7 years postmenpopausal with the absence of vaginal bleeding for at least 1 year
* ≥ 24 in mini mental state examination
* not suffering from psychiatric distress as assessed using GHQ28 questionnaire

Exclusion Criteria:

* surgically induced menopause
* habitual consumers of soys foods (> 2 serves/week)
* currently using hormone therapy
* currently on isoflavone supplements
* antibiotics use within last 3 months
* use of psychoactive medication
* history of CVD, cancer, diabetes, thyroid, renal or kidney disease, alcohol or drug abuse
* red-green colour blindness

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive function | Change at Week 12 from baseline
  Assessed using the computerised Cambridge Neuropsychological Test Automated Battery (CANTAB)

SECONDARY OUTCOMES:
Change in Menopausal symptoms | Change at Week 12 from baseline
  Greene's Climacteric scale, a 21 item scale measuring menopausal symptoms, including psychological, somatic and vasomotor symptoms, it is scored on a scale from 0-63, with higher scores indicating greater severity of symptoms.
Change in Quality of Life | Change at Week 12 from baseline
  Control, Autonomy, Self-realisation and Pleasure (CASP-19). CASP 19 is a measure of quality of life, it has 19 questions comprising 4 subscales assessing control, autonomy, self-realisation and pleasure, scored from 0-3, subscales range from 0-12 and 0-15, with higher scores indicating higher quality of life.
Change in Mood | Change at Week 12 from baseline
  Positive and Negative Affect Schedule (PANAS), a 20 item questionnaire assessing positive and negative mood, a score is calculated for each of these and range from 1-50, with higher scores indicating greater presence of the mood.
Change in Stress | Change at Week 12 from baseline
  Perceived stress scale, a 14 item questionnaire measuring global stress levels with a higher score indicating greater psychological distress. Scores can range from 0-52.
Change in Coping | Change at Week 12 from baseline
  COPE Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No